CLINICAL TRIAL: NCT02880462
Title: Phase 2 Study of the Effect of add-on Sulforaphane in Treatment of Schizophrenia
Brief Title: A 6-month Study to Evaluate Sulforaphane add-on Effects in Treatment of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Stanley-Sulforaphane
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; sulforaphane
MeSH Terms: conditions — Schizophrenia | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and researchers are blind to treatment allocation (double-blind). An independent researcher developed the computer-generated randomization plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose sulforaphane (Active Comparator): The goal of the study is to investigate whether adding high doses of sulforaphane will benefit the clinical symptoms and cognitive function in individuals who have schizophrenia.
  Interventions: Dietary Supplement: sulforaphane
- low dose sulforaphane (Active Comparator): The goal of the study is to investigate whether adding low doses of sulforaphane will benefit the clinical symptoms and cognitive function in individuals who have schizophrenia.
  Interventions: Dietary Supplement: sulforaphane
- placebo (Placebo Comparator): The purpose of including placebo is to judge if the outcome is related to the study medication rather than other reasons.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: sulforaphane — Sulforaphane is a compound that can be extracted from broccoli, Brussel sprouts, cabbage, and other cruciferous plants.
  Other Names: Nutramax
  Arms: high dose sulforaphane; low dose sulforaphane
Other: placebo — Placebo is made of starch
  Arms: placebo

SUMMARY:
The goal of the study is to investigate whether adding different doses of sulforaphane will benefit the clinical symptoms and cognitive function in individuals who have schizophrenia.

This study will compare the sulforaphane with placebo. There is a thirty percent change (less than half) of receiving the placebo. The purpose of including placebo is to judge if the outcome is related to the study medication rather than other reasons.

DETAILED DESCRIPTION:
This study will be carried out in six mental health institutes in China and total of 180 patients with first-episode or early onset schizophrenia will be enrolled into the study. The mental health institute at the Second Xiangya Hospital, Central South University.

Individuals who participate in the study will be followed for 24 weeks. The changes in clinical symptoms and neurocognitive function will be assessed from baseline (week-2) to week-6 (acute phase), and week-12 to week-24 (maintenance phase).

ELIGIBILITY:
Inclusion Criteria:

1. Meet The Diagnostic and Statistical Manual (DSM-V) diagnostic criteria for schizophrenia
2. First onset or duration of illness less than 3 years with current symptoms exacerbation
3. Hospitalized in an acute episode (first hospitalization), or subsequent hospitalization or acute relapse)
4. Male and female with aged 18 to 50 years
5. PANSS total >=75 at 2 weeks. .
6. Signed the study consent for participation

Exclusion Criteria:

1. having history of substance dependence or abuse or whose symptoms are caused by the other diagnosable mental disorders;
2. having history of traumatic brain injury, seizures or other known neurological or organic diseases of the central nervous system;
3. taking antidepressants, stimulants, mood stabilizer or accepts electricity shock treatment;
4. having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be manage in an inpatient setting;
5. the routine blood tests showing abnormal renal, liver function or other metabolic results .
6. pregnant or lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Cognitive improvement assessed using the MATRICS Consensus Cognitive Battery (MCCB) composite score | 24 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure.

SECONDARY OUTCOMES:
side effects by SAFTEE | 24 weeks
  The investigators will evaluate side effect by The Systematic Assessment for Treatment Emergent Events (SAFTEE).
side effects by AIMS | 24 weeks
  The investigators will evaluate side effect by Abnormal Involuntary Movement Scale (AIMS)
side effects by BAS | 24 weeks
  The investigators will evaluate side effect by Barnes Akathisia Rating Scale (BAS).
side effects by SAS | 24 weeks
  The investigators will evaluate side effect bySimpson-Angus Scale (SAS).
Change of clinical symptoms by PANSS | 24 weeks
  The change of Positive And Negative Syndrome Scale (PANSS) total, positive and negative symptoms before and after treatment at different follow up point
Change of clinical symptoms of CGI | 24 weeks
  The change of Clinical Global Impression (CGI) before and after treatment at different follow up point

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, M.D Ph.D, Principal Investigator — Central South University; Renrong Wu, M.D Ph.D, Principal Investigator — Central South University; Jingping Zhao, M.D Ph.D, Study Chair — Central South University; Hua Jin, M.D Ph.D, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Selley ML. Increased (E)-4-hydroxy-2-nonenal and asymmetric dimethylarginine concentrations and decreased nitric oxide concentrations in the plasma of patients with major depression. J Affect Disord. 2004 Jun;80(2-3):249-56. doi: 10.1016/S0165-0327(03)00135-6. PMID 15207938
- [Background] Bitanihirwe BK, Woo TU. Oxidative stress in schizophrenia: an integrated approach. Neurosci Biobehav Rev. 2011 Jan;35(3):878-93. doi: 10.1016/j.neubiorev.2010.10.008. Epub 2010 Oct 23. PMID 20974172